CLINICAL TRIAL: NCT03670914
Title: Diagnosis of Sleep-Related Respiratory Disorders in Patients With Narcotic Medications
Acronym: WP-NARC001
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: Due to the recent COVID-19 surge the majority of our staff was pulled from sleep care to inpatient care. Thus, we have had to temporarily pause in-lab studies until our staff returns. We hope to proceed with recruitment as soon as possible.
Sponsor: Kaiser Permanente (Other)
Responsible Party: Principal Investigator, Dennis Hwang, MD, Department Medical Director, Kaiser Permanente
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: WatchPAT200-NARC001
Record Dates: First submitted 2018-09-12; First posted 2018-09-14 (Actual); Last update posted 2022-07-06 (Actual); Status verified 2022-07

CONDITIONS: Narcotic Use; Central Sleep Apnea
Keywords: Sleep Disorder Breathing; Central Sleep Apnea; Narcotics; Home Sleep Apnea Testing Device; WatchPAT 200; In-Lab Polysomnography; Comparison; Accuracy; Efficacy
MeSH Terms: conditions — Sleep Apnea, Central

STUDY DESIGN:
Intervention Model Description: This is a prospective single cohort study that will evaluate the efficacy of the WatchPAT200 device by comparing it to an in-lab polysomnography.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- WatchPAT 200 and In-Lab Study (Experimental): Patients who are referred to the sleep center for an overnight study that are narcotic users will be offered to the opportunity to participate in the study. Patients who fulfill the inclusion exclusion criteria and have given informed consent will undergo a standard in-lab polysomnography while simultaneously wearing the WatchPAT200 device.
  Interventions: Diagnostic Test: WatchPAT 200

INTERVENTIONS:
Diagnostic Test: WatchPAT 200 — The WatchPAT200 device has been approved by the Food and Drug Administration (FDA) for testing sleep related disorders in patients ages 17 and older. They are widely used with thousands of studies performed in the United States to validate the devices accuracy and efficacy. It is also routinely used in many other countries. The devices are not currently being used for patients who are currently taking narcotic medications at Kaiser Permanente. Therefore, we are asking patients to simultaneously wear this device during an in-lab study, so we can test how effective and accurate the WatchPAT 200 is in diagnosing sleep breathing disorders in patients on narcotic medications.

SUMMARY:
The present study is a prospective, single cohort study involving patients on narcotic medications, undergoing overnight sleep studies in the clinical sleep laboratory. The main hypothesis for the study is that the the frequency of sleep respiratory events (including central apneas) identified by a home sleep apnea test (HSAT) device (WatchPAT200U (wp200U) with centrals; Itamar Medical Ltd.) will significantly correlate with in-lab polysomnography (gold standard).

DETAILED DESCRIPTION:
Background

Opioid use in the United States has escalated on an unprecedented scale since 1997, when the American Academy of Pain Medicine and the American Pain Society issued a statement declaring that respiratory depression typical to opioid use is a significant concern. The Trends and Risks of Opioid Use for Pain (TROUP) study demonstrated a broad-based increase in the use of potent opioids in publicly and privately insured enrollees between 2000 and 2005. Their findings suggest a significant liberalization in opioid use for non-cancer pain that is not limited to one geographic region or socioeconomic group.

Chronic use of opioid medication' (i.e., longer than 6 months) predisposes patients to the development of an irregular breathing pattern with central apneas during sleep, best characterized as Biot's respiration, ataxic breathing. Ataxic breathing is characterized by a breathing pattern in which there are groups of similar sized breaths alternating with regular periods of central apnea.

The WatchPAT HSAT device and polysomnography are both standard diagnostic tests for sleep disordered breathing, in particular for obstructive sleep apnea. However, the WatchPAT has never been validated in regards to its diagnostic accuracy pertaining to narcotic-induced central apneas.

This study has important implications to the medical field and patients for the following reasons:

1. Narcotic induced central sleep apnea is a marker for respiratory suppression and is thought to increase the risk of respiratory failure, hospital admission, and death. Validating the accuracy and reliability of WatchPAT is a more cost-efficient and accessible test than polysomnography and thus improves patient access and better identification of this problem in patients at risk. If the accuracy is validated, this would potentially benefit our patients by allowing those patients to be tested at home (more convenient), require less wait time (access for full polysomnography (PSG) is prolonged), and reduce healthcare costs (PSG is about 10-fold more expensive that home sleep apnea testing).
2. WatchPAT is one of the most commonly used HSAT devices. Thus, validating its technology has significant implications in sleep testing workflow throughout the nation.

Study Design

Recruitment

Patients who are referred to the sleep center, clinically identified to be at risk for narcotic-induced central sleep apnea and triaged to polysomnography testing will be eligible for recruitment. Investigators will perform a preliminary eligibility chart review and will contact potentially eligible patients by telephone to ask patients whether they would be interested in participating in a research study. Investigators will confirm eligibility, review the study protocol and informed consent utilizing an Institutional Review Board (IRB) approved telephone script for those who are interested in participating. Patients who have expressed verbal consent will be mailed or emailed a blank copy of the informed consent form (ICF) to allow for review prior to the sleep study. For those that elect for the ICF to be emailed, a blank ICF will be emailed from either Health Connect (via KP.org) or an internal Kaiser Permanente (KP) Outlook email utilizing an IRB approved email script. The patient will be provided with contact information for any questions during the time in between receiving the ICF and night of their sleep study. The phone recruitment process with the patient will generally occur as follows:

1. During each investigator's standard review of the chart of patients already scheduled for polysomnography and determine their risk of narcotic induced central sleep apnea based on the investigator's (physician) clinical judgment.
2. In the event that either investigator identifies an eligible patient, he will then prepare the eligibility form for the subject and contact the patient.
3. During the recruitment phone call with the patient who is eligible for the study, the investigator will follow the proposed telephone script to a review of the protocol, study risks, study procedures, and final consenting plan. At the moment of the phone conversation the investigator will give the patient the opportunity to ask questions. The investigator will attempt 3 recruitment phone calls. If he is unable to contact the patient after 3 tries (including voicemails and direct contact messages), he will consider that patient a recruitment fail.
4. Once the patient expresses their verbal consent for the study and documented in Health Connect, the investigator will ask if the patient has any finger deformity, which disqualifies the patient from the study, and confirm the patient takes narcotic medication at least 4 nights/week. Once those inclusion/exclusion criteria are confirmed and communicated, the investigator will finalize the eligibility form by personally signing and dating, and then the investigator or designee will either mail or email the patient a blank copy of the ICF within 2 business days, to allow for review of the ICF prior to the sleep study visit. For those patients electing for the ICF to be emailed, the investigator or designee will email the blank ICF from their internal Kaiser Permanente Outlook email. The patient will be provided with contact information for any questions during the time between them receiving the ICF and the sleep study visit.

In-Person Consenting Process

Once the investigator receives a verbal consent from the patient, the investigator will inform the Research Associate, the designated sleep technician and/or department administrator that is scheduled to work at the Sleep Lab the night the patient is scheduled, about the potential subject. The subject will be asked to be in the sleep lab at the usual scheduled time (overall, per standard of care, the sleep study will end at 6:00 am the following morning). The in-person consenting process with the patient will generally occur as follows:

1. The Sleep Lab Technician or Department Administrator, who completed the appropriate clinical trials required training (i.e. Health Insurance Portability and Accountability Act (HIPAA), IRB Standard Operating Procedure 502 (SOP 502), and Collaborative Institutional Training Initiative Good Clinical Practice (CITI GCP)) along with protocol training, to obtain consent and are designated by the PI, will obtain a written informed consent from the patient by reviewing the IRB-approved ICF. The patient will be given time to review the ICF to signing the form in accordance to GCP and the regulatory, legal requirements.
2. The patient will be given a copy of the signed ICF by the person obtaining consent (e.g. Sleep Technician, Department Administrator) after a review that the documents were properly signed.
3. The in-person consenting process will also be documented in the subject's records by the person obtaining consent (e.g. Sleep Technician, Department Administrator)

Consenting Process Training and Supervision Study site staff will be trained by the Investigator and Research Associate on the two part consenting process in the following way: (1) investigators will be trained for recruitment with verbal consent via phone and (2) sleep technicians and department administrators will be trained for in-person consenting. The supervision of the two-part consenting process is delegated to the Primary Investigator and Research Associate. The primary investigator and/or Research Associate will be present during the first subject in-person consenting for each Sleep Technician and Department Administrator to ensure that they understand the requirements.

Patients who have consented will undergo an in-lab PSG while simultaneously wearing the WatchPAT200. The WatchPAT200 is a wrist device which contains a pulse oximeter probe and an external snoring/body position (SBP) sensor (SBP is attached to the subject's chest just under the sternal notch). Authorized and trained investigators/ evening sleep technicians will be responsible for setting up PSG and WatchPAT200 equipment on all research patients. Technicians will also be responsible for attaching a synchronization cable from the WatchPAT200 device to a PSG auxiliary Direct Current (DC) channel to sync data for 15 minutes at the start and end of the sleep study. The technicians will only score PSG data and will not have access to the WatchPAT200 data.

During the day, a trained investigator or daytime technician will be responsible for downloading the WatchPAT200 data and setting up the device for the next research patient.

Participants will not be compensated for this study, although co-payment for the in-lab PSG will be waived and participants will not have to pay for the additional WatchPAT200 testing.

Patient baseline characteristics (gender, age, BMI, Epworth Sleepiness Scale (ESS), etc.) will be acquired from the patient themselves and/or from the patient's medical chart. The data obtained by the WatchPAT200 will be analyzed automatically by the WatchPAT200 software (zzzPAT) and will be compared to the PSG's manual scoring. Variability in the following data will be assessed and analyzed between PSG and WatchPAT200:

1. Respiratory and oximetry data (Apnea-hypopnea index, oxygen disturbance index, respiratory disturbance index, oxygen saturation, central apnea index, central hypopnea index, total central index, periodic breathing, etc.)
2. Sleep position and staging data (supine time, Rapid Eye Movement (REM) time, sleep time, etc.)
3. Sleep-wake data (analyzed time, sleep time, sleep efficiency, etc.)

ELIGIBILITY:
Inclusion Criteria

* Kaiser Permanente member
* Patient is able to read, understand and sign the informed consent form.
* Subject on current narcotic prescription with of at least 4 nights/week (subject will be asked on night of PSG if they took narcotic medication and specific medication taken)

Exclusion Criteria

* Finger deformity that precludes adequate sensor appliance
* Use of one of the following medications: alpha blockers, short acting nitrates (less than 3 hours before the study)
* Patients that are oxygen dependent
* Patients with Chronic Obstructive Pulmonary Disease (COPD) with FEV1 <70%, obesity hypoventilation syndrome, neuromuscular weakness

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2019-08-08 (Actual); Primary Completion 2023-07 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Accuracy of Central Sleep Apnea Events | 1 year
  Compare the efficacy of the WatchPAT200 in detecting narcotic based central respiratory events to the manual scoring of the in-lab polysomnography that serves as a "gold standard".
Accuracy of Other Various Sleep Metrics | 1 year
  Compare the efficacy of the WatchPAT200 in detecting narcotic based oxygen, body position, and sleep-wake events to the in-lab polysomnography.

CONTACTS AND LOCATIONS:
Overall Officials: Dennis Hwang, MD, Principal Investigator — Kaiser Permanente Fontana Medical Sleep Center
Locations (1):
- Sleep Center; San Bernardino County Medical Center, Kaiser Permanente, Fontana, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chou R, Clark E, Helfand M. Comparative efficacy and safety of long-acting oral opioids for chronic non-cancer pain: a systematic review. J Pain Symptom Manage. 2003 Nov;26(5):1026-48. doi: 10.1016/j.jpainsymman.2003.03.003. PMID 14585554
- [Background] Sullivan MD, Edlund MJ, Fan MY, DeVries A, Braden JB, Martin BC. Trends in use of opioids for non-cancer pain conditions 2000-2005 in commercial and Medicaid insurance plans: the TROUP study. Pain. 2008 Aug 31;138(2):440-449. doi: 10.1016/j.pain.2008.04.027. Epub 2008 Jun 10. PMID 18547726
- [Background] Walker JM, Farney RJ, Rhondeau SM, Boyle KM, Valentine K, Cloward TV, Shilling KC. Chronic opioid use is a risk factor for the development of central sleep apnea and ataxic breathing. J Clin Sleep Med. 2007 Aug 15;3(5):455-61. PMID 17803007